CLINICAL TRIAL: NCT05503121
Title: Investigation of the Relationship Between Biomarkers and Biomechanical Properties in Individuals With Nonspecific Low Back Pain
Brief Title: Relationship Between Biomarkers and Biomechanical in Nonspecific Low Back Pain
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Istinye University (Other)
Collaborators: The Scientific and Technological Research Council of Turkey (Other)
Responsible Party: Sponsor
Other Study IDs: 3/2022.K-65
Record Dates: First submitted 2022-08-10; First posted 2022-08-16 (Actual); Last update posted 2022-08-16 (Actual); Status verified 2022-08

CONDITIONS: Low Back Pain
Keywords: Biomarker; Biomechanic; Nonspecific low back pain; 3D motion analysis system; sEMG
MeSH Terms: conditions — Low Back Pain

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Study Group: The volunteer group planned to be included in the study will consist of individuals diagnosed with Nonspecific Low Back Pain who applied to Istinye University Physiotherapy and Rehabilitation Application and Research Center (Isu Fizyotem).
  21 volunteers with low back pain will be included in the study.
  Interventions: Diagnostic Test: 3D motion analysis, muscle activation, biomarker analysis
- Contol Group: The control group will consist of healthy individuals. 21 healty volunteers will be included in the study.
  Interventions: Diagnostic Test: 3D motion analysis, muscle activation, biomarker analysis

INTERVENTIONS:
Diagnostic Test: 3D motion analysis, muscle activation, biomarker analysis — Participants with nonspesific low back pain and control group will be analysed with 3D motion analysis sistem, sEMG and will be checked the biomarkers. Then the data will be compared.

SUMMARY:
Nonspecific low back pain is one of the most common health problems today. Although it is encountered so frequently, the relationships between the symptoms of patients who complain of low back pain have not been fully explained.

With pain, changes occur in the body of individuals. When the blood values of individuals are examined, changes are observed in their biomarkers. Two of these biomarkers are anti-inflammatory and pro-inflammatory biomarkers. These two biomarkers indicate that there is an inflammation in the body. Inflammation can cause pain. Pain also prevents individuals from performing their movements correctly and can cause individuals to make biomechanical changes in their bodies that will make them feel less pain. Clinicians and physiotherapists treat symptoms for pain, patients' pain starts again or does not go away at all because the underlying problem is not fully understood and resolved.

Biomechanical features that can be explained as muscle activation and joint movements can be defined as the lowest unit of functional movement. These movements combine to form functions. When we search for functionality in the literature, we see that the functionality increases with the decrease of inflammation. Functions performed in a different way than normal due to pain and changes in these functions may or may not be at an observable level. For this reason, the biomechanical changes of individuals with pain will be analyzed with a more detailed and objective measurement system.

The three-dimensional motion analysis system and muscle activation measuring devices to be used in this study are devices that can make the most accurate and precise measurement and allow us to examine the lowest unit of motion. This study will go to the basis of the movement and understand the problems there and will contribute to the production of permanent solutions in future studies.

Pain and biomarkers and pain and biomechanical properties were evaluated separately in the studies, no study was found that examined biomechanical properties and biomarkers together. The aim of the project is to examine the relationship between inflammation and biomechanical properties. At the end of the project, the relationship between inflammation and biomechanical changes in low back pain will be demonstrated objectively, and it is anticipated that new treatment strategies can be developed for nonspecific low back pain.

ELIGIBILITY:
Inclusion Criteria:

* Nonspecific low back pain diagnosed by a physical therapy and rehabilitation specialist,
* For participants with pain, those who defined their pain on a scale of 3-7 on VAS,
* Individuals between the ages of 18-45 who have had pain in the lumbar region for at least 3 months,
* Those who do not have an infectious condition for any other reason (gum infection, metabolic diseases, viral infections, etc.) will be included in the study.

Exclusion Criteria:

* Diagnosed with disc herniation,
* diagnosed with scoliosis,
* Lumbal spine surgery or lumbar spine trauma,
* Those with a history of spine infection, tumor, osteoporosis, structural deformity, cauda equina syndrome, radicular syndrome,
* Those who participated in the period 1 week before and 1 week after the menstrual cycle,
* Diagnosed with rheumatic disease,
* Individuals with difficulty in cooperation and
* Individuals who received physical therapy within 3 months will not be included in the study.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Individuals between the ages of 18-45 who have had nonspecific low back pain.
Sampling Method: Non-Probability Sample
Enrollment: 42 (Estimated)
Dates: Start 2022-09-01 (Estimated); Primary Completion 2022-11-20 (Estimated); Study Completion 2023-02-01 (Estimated)

PRIMARY OUTCOMES:
Motion analysis | baseline
  Noraxon MyoMotion 3D motion analysis system will be used. Inertial measurement unit (IMU) are placed on any body segment with elastic fixation straps.
  The sensors will be placed in the spinal processes of Thoracic 12, Lumbar 3 and Sacral 2 with adjustable straps. The participant is asked to stand while placing the sensors. T12 level is found by palpating the spinal processes of the spines. Sacral 2 spinal process is palpated from line between right and left posterior superior spina iliaca. efore each measurement, the IMU sensors will be calibrated for body position. Data collected with a sampling frequency of 200 Hz will be recorded. A laptop camera will be used as a camera during the measurements.
Muscle activation | baseline
  Noraxon MyoMuscle system will be used. The MyoMuscle system processes the signals sent by superficial electromyography (sEMG) electrodes placed on the participants' body. The electrodes used in sEMG measurement are Ag/AgC superficial electrodes. In the EMG analysis, 2 muscle groups will be evaluated, and the electrodes will be placed bilaterally.
  Lumbal erector spines: Electrodes is placed 3 cm lateral to the spinal process of the fourth lumbar spine.
  Obliquus internus: The electrode is placed 2 cm medial to the anterior superior iliac spine.
  The signals of muscle movements of the electrode-placed muscles during standing up from sitting will be measured.
  TeleMyo DTS will be used to collect EMG data. Collected data will be filtered by MyoResearch XP 1.72 software.
Short Form McGill Pain Questionnaire | baseline
  The McGill Pain Questionnaire consists of a total of 15 descriptive words. Of the 15 words used to evaluate the dimensions of pain, 11 are used to evaluate the sensory and 4 are used to evaluate the affective dimensions of pain. Pain intensity is scored by the patient as 0=absent, 1=mild, 2=moderate, 3=severe. Total scores are scored at three levels: sensory, affective, and total (sensory+affective). The Short Form McGill questionnaire has a visual analog scale used to assess the severity of pain and a 6-point Likert scale. In the Likert scale of SF- McGill index, 0 = no pain, 1 = mild, 2 = bothersome, 3 = distressing, 4 = awful, 5 = excruciating pain.
Analysis of Inflammatory Markers (Interleukin-1Beta, Tumor Necrosis Factor Alpha, Interleukin-6, Interleukin-2, Interleukin-8, Interleukin-10 ) | baseline
  Changes between individuals with low back pain and healthy individuals.

IPD SHARING:
Plan to Share IPD: No